CLINICAL TRIAL: NCT06349044
Title: A Randomized, Multicenter Phase II Basket Study of Hypofractionated Radiotherapy/Stereotactic Body Radiotherapy Followed by Immunotherapy-Based Systemic Therapy +/- L. Rhamnosus M9 for the First-Line Treatment of Advanced Digestive System Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ji Zhu, Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BASIMA
Record Dates: First submitted 2024-03-21; First posted 2024-04-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Her-2 Negative Adenocarcinoma of the Gastro-oesophageal Junction/Gastric Adenocarcinoma; Hepatocellular Carcinoma; Biliary Tract Carcinoma; Colorectal Adenocarcinoma
Keywords: radiotherapy; immunotherapy; L. rhamnosus M9
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — spartalizumab; Oxaliplatin; Capecitabine; Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- ARM A:Her-2 negative adenocarcinoma of the gastroesophageal junction/gastric adenocarcinoma (Experimental): patients will receive Probio-M9 ,RT followed by Immunotherapy-Based Systemic Therapy
  Interventions: Radiation: Hypofractionated radiotherapy/SBRT（5-10Gy/fx，3-5 fx）; Drug: Anti-PD-1 monoclonal antibody; Drug: Oxaliplatin and Capecitabine
- ARM A*:Her-2 negative adenocarcinoma of the gastroesophageal junction/gastric adenocarcinoma (Placebo Comparator): patients will receive placebo ,RT followed by Immunotherapy-Based Systemic Therapy
  Interventions: Radiation: Hypofractionated radiotherapy/SBRT（5-10Gy/fx，3-5 fx）; Drug: Anti-PD-1 monoclonal antibody; Drug: Oxaliplatin and Capecitabine
- ARM B: Liver adenocarcinoma (Experimental): patients will receive Probio-M9 ,RT followed by Immunotherapy-Based Systemic Therapy
  Interventions: Radiation: Hypofractionated radiotherapy/SBRT（5-10Gy/fx，3-5 fx）; Drug: Anti-PD-1 monoclonal antibody; Drug: Anti-VEGF 15mg/kg
- ARM B*: Liver adenocarcinoma (Placebo Comparator): patients will receive placebo ,RT followed by Immunotherapy-Based Systemic Therapy
  Interventions: Radiation: Hypofractionated radiotherapy/SBRT（5-10Gy/fx，3-5 fx）; Drug: Anti-PD-1 monoclonal antibody; Drug: Anti-VEGF 15mg/kg
- ARM C: Malignant tumors of the biliary system (Experimental): patients will receive Probio-M9 ,RT followed by Immunotherapy-Based Systemic Therapy
  Interventions: Radiation: Hypofractionated radiotherapy/SBRT（5-10Gy/fx，3-5 fx）; Drug: Anti-PD-1 monoclonal antibody; Drug: Gemcitabine and Cisplatin
- ARM C*: Malignant tumors of the biliary system (Placebo Comparator): patients will receive placebo ,RT followed by Immunotherapy-Based Systemic Therapy
  Interventions: Radiation: Hypofractionated radiotherapy/SBRT（5-10Gy/fx，3-5 fx）; Drug: Anti-PD-1 monoclonal antibody; Drug: Gemcitabine and Cisplatin
- ARM D:Colorectal cancer (Experimental): patients will receive Probio-M9 ,RT followed by Immunotherapy-Based Systemic Therapy
  Interventions: Radiation: Hypofractionated radiotherapy/SBRT（5-10Gy/fx，3-5 fx）; Drug: Anti-PD-1 monoclonal antibody; Drug: Oxaliplatin and Capecitabine; Drug: Anti-VEGF 7.5mg/kg
- ARM D*:Colorectal cancer (Placebo Comparator): patients will receive placebo ,RT followed by Immunotherapy-Based Systemic Therapy
  Interventions: Radiation: Hypofractionated radiotherapy/SBRT（5-10Gy/fx，3-5 fx）; Drug: Anti-PD-1 monoclonal antibody; Drug: Oxaliplatin and Capecitabine; Drug: Anti-VEGF 7.5mg/kg

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy/SBRT（5-10Gy/fx，3-5 fx） — RT: one primary or metastatic focus was selected for hypofractionated radiotherapy/SBRT (5-10 Gy/fx, 3-5 fx) in each round, the target area included only the GTV of the visible tumor lesion, and the GTV was expanded by 5-10 mm to generate the PTV, and the prophylactic lymphatic drainage area could not be irradiated.
Drug: Anti-PD-1 monoclonal antibody — Sintilimab 200mg d1 iv q3w
Drug: Oxaliplatin and Capecitabine — Oxaliplatin130mg/m2 d1 iv；Capecitabine1000mg/m2 d1-d14
  Arms: ARM A*:Her-2 negative adenocarcinoma of the gastroesophageal junction/gastric adenocarcinoma; ARM A:Her-2 negative adenocarcinoma of the gastroesophageal junction/gastric adenocarcinoma; ARM D*:Colorectal cancer; ARM D:Colorectal cancer
Drug: Anti-VEGF 15mg/kg — Bevacizumab 15mg/kg d1 iv q3w
  Arms: ARM B*: Liver adenocarcinoma; ARM B: Liver adenocarcinoma
Drug: Anti-VEGF 7.5mg/kg — Bevacizumab 7.5mg/kg d1 iv q3w
  Arms: ARM D*:Colorectal cancer; ARM D:Colorectal cancer
Drug: Gemcitabine and Cisplatin — Gemcitabine1000mg/m2 d1 d8 iv；Cisplatin 25mg/m2 d1 d8 iv q3w
  Arms: ARM C*: Malignant tumors of the biliary system; ARM C: Malignant tumors of the biliary system

SUMMARY:
Based on the interaction between radiation therapy and immunotherapy and the potential potentiation of Probio-M9 for the treatment of ICIs, this study is planned to design an integrated treatment protocol for the first-line treatment of advanced gastrointestinal tumors through the use of macrofractionated radiotherapy as a means of immune activation, combined with the synergistic effect of Probio-M9 microbial agents and PD-1 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* histopathologically confirmed diagnosis of malignant tumors of the gastrointestinal tract (including Her-2 negative adenocarcinoma of the gastroesophageal junction/gastric adenocarcinoma, hepatocellular carcinoma, malignant tumors of the biliary system, colorectal cancer);
* advanced patients evaluated as initially non-operable resectable who have not received any antitumor therapy;
* have at least one measurable or evaluable lesion according to RECIST v1.1 criteria in addition to the primary lesion, with non-operable resectable lymph node metastases to the liver, lung, bone, pelvis, retroperitoneum and/or superficial sites (except for brain metastases), as evaluated by discussion in the framework of the MDT
* age 18-75 years;
* ECOG score of 0-1;
* be able to accept the treatment regimen during the study;
* sign a written informed consent.

Exclusion Criteria:

* a history of uncontrolled epilepsy, central nervous system disease, or psychiatric disorder of clinical severity that, in the judgment of the investigator, may preclude the signing of an informed consent form or interfere with the patient's adherence to oral medication;
* prior immunotherapy for any indication or a history of severe hypersensitivity reactions to other monoclonal antibodies;
* clinically significant (i.e., active) cardiac disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) class II or worse congestive heart failure or severe arrhythmias requiring pharmacologic intervention, or history of myocardial infarction within the last 12 months;
* organ transplantation requiring immunosuppressive therapy;
* a history of other malignant disease within the last five years;
* persons with severe uncontrolled recurrent infections, or other severe uncontrolled concomitant diseases;
* Subjects whose baseline blood routine and biochemical indexes do not meet the following criteria: hemoglobin ≥80g/L; absolute neutrophil count (ANC) ≥1.5×10^9/L; platelets ≥100×10^9/L; ALT, AST ≤2.5 times the upper limit of normal; ALP ≤2.5 times the upper limit of normal; serum total bilirubin <1.5 times the upper limit of normal; serum creatinine <1 times the upper limit of normal; and serum creatinine <1 times the upper limit of normal. times the upper limit of normal;
* the patient currently has active gastrointestinal diseases such as active gastric and duodenal ulcers, ulcerative colitis, or active bleeding from unresected tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by the investigator;
* persons with active bleeding or bleeding tendencies;
* women who are pregnant or breastfeeding;
* allergy to any of the study drug ingredients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | ORR will be assessed 2 months after radiotherapy
  for off-target lesions of radiotherapy

SECONDARY OUTCOMES:
ORR | ORR will be assessed 2 months after radiotherapy
  irradiated lesion
adverse effects rate | From date of randomization until the date of death from any cause, assessed up to 5 years ]
  CTC 4.0
Qol | From date of randomization until the date of death from any cause, assessed up to 10 years]
  EORTC-C30
PFS | From the date of randomization to the date when progress was first recorded,assessed up to 36 months.
  Rate of 3 year disease free survival
OS | From date of randomization until the date of death from any cause, assessed up to 36 months
  Rate of 3 year overall survival
Qol | From date of randomization until the date of death from any cause, assessed up to 10 years]
  EQ-5D

CONTACTS AND LOCATIONS:
Locations (1):
- Zhengjiang Cancer Hospital, Hangzhou, Zhejiang, China